CLINICAL TRIAL: NCT05311501
Title: Impact of Non-surgical Periodontal Therapy in the Management of Plaque Psoriasis. A Randomised Controlled Trial.
Brief Title: Impact of Non-surgical Periodontal Therapy in the Management of Plaque Psoriasis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Simone Grandini, Full Professor, University of Siena
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TPSO001
Record Dates: First submitted 2022-03-16; First posted 2022-04-05 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Psoriasis Vulgaris; Psoriasis; Periodontitis
MeSH Terms: conditions — Psoriasis; Periodontitis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate periodontal treatment (Experimental): Right after the execution of a complete periodontal chart, non-surgical periodontal treatment (NST) was performed, according to the most recent clinical guidelines. NST was performed by removing supra and subgingival calculus and using both ultrasonic and manual instruments. Oral Hygiene Instructions (OHI) were provided throughout the experimental period.
  Interventions: Other: Non-surgical periodontal treatment
- Delayed Periodontal treatment (No Intervention): Right after the execution of a complete periodontal chart, the patient is informed regarding their group allocation, according to which they are asked to delay NST for 10 weeks. 10 weeks after baseline examination, NST was performed according to the most recent clinical guidelines. NST was performed by removing supra and subgingival calculus and using both ultrasonic and manual instruments.

INTERVENTIONS:
Other: Non-surgical periodontal treatment — Non-Surgical periodontal Treatment was performed by removing supra and subgingival calculus and using both ultrasonic and manual instruments. Oral Hygiene Instructions (OHI) were provided throughout the experimental period. Local anesthesia was performed only when needed.
  Arms: Immediate periodontal treatment

SUMMARY:
Both periodontitis and plaque psoriasis are non communicable chronic inflammatory diseases. They share genetic polymorphysms (IL-1, IL-6 e TNFalfa) and risk factors (smoking, diabetes, obesity), as well as a great resemblance in terms of pathophysiological pathways. In fact, they are both characterized by an hyperactivation of the innate immune response which induces an excessive production of cytokines such as IL-17/TNFalfa. While non-surgical periodontal therapy consists in the mechanical removal of supra and subgingival calculus, psoriasis treatment involves the administration of either systemic or biologic drugs. Evidence is scarce regarding the effectiveness of non-surgical periodontal therapy in ameliorating the clinical outcomes of plaque psoriasis. The biological plausibility relies on the important reduction of systemic inflammation caused by periodontal treatment, which could ameliorate psoriasis phenotype.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of plaque psoriasis;
* diagnosis of untreated periodontitis;
* presence of at least 20 teeth;
* age between 18 and 70 years;
* ability and willingness to give informed consent.

Exclusion Criteria:

* inability of unwillingness to give informed consent;
* patients undergoing periodontal treatment within the last 6 months;
* patients undergoing immunosuppressive treatments for other systemic diseases;
* pregnancy or lactation;
* pts undergoing antibiotic therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
PASI (Psoriasis Area and Severity Index)- Baseline | PASI was registered at baseline.
  A representative area of psoriasis is selected for each body region (head and neck, upper and lower limbs, trunk). The intensity of redness, thickness, and scaling of the psoriasis is assessed as none (0), mild (1), moderate (2), severe (3), or very severe (4). The three intensity scores are added up for each of the four body regions to give subtotals A1, A2, A3, A4.
  Each subtotal is multiplied by the body surface area represented by that region. The higher the score, the worse psoriasis severity.
PASI (Psoriasis Area and Severity Index)- 10 weeks | PASI was registered 10 weeks after baseline.
  A representative area of psoriasis is selected for each body region (head and neck, upper and lower limbs, trunk). The intensity of redness, thickness, and scaling of the psoriasis is assessed as none (0), mild (1), moderate (2), severe (3), or very severe (4). The three intensity scores are added up for each of the four body regions to give subtotals A1, A2, A3, A4.
  Each subtotal is multiplied by the body surface area represented by that region. The higher the score, the worse psoriasis severity.

SECONDARY OUTCOMES:
Body Surface Area (BSA)- Baseline | BSA was registered at baseline.
  BSA is calculated as the extent to which the body is affected by psoriasis. The score ranges between 0 and 100; the higher the score, the worse psoriasis severity.
Body Surface Area (BSA)- 10 weeks | BSA was registered 10 weeks after baseline.
  BSA is calculated as the extent to which the body is affected by psoriasis. The score ranges between 0 and 100; the higher the score, the worse psoriasis severity.

OTHER OUTCOMES:
Salivary Concentration of miRNAs- Baseline | Salivary Concentration of miRNAs was registered at baseline.
  The salivary concentration of specific miRNAS involved in both psoriasis and periodontitis (miRNA146a, miRNA223, miRNA21, miRNA155) was detected. The higher the concentration, the worse the severity of both periodontitis and psoriasis.
Salivary Concentration of miRNAs- 10 weeks | Salivary Concentration of miRNAs was registered 10 weeks after baseline.
  The salivary concentration of specific miRNAS involved in both psoriasis and periodontitis (miRNA146a, miRNA223, miRNA21, miRNA155) was detected. The higher the concentration, the worse the severity of both periodontitis and psoriasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Senese, Siena, Italy

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be made available upon reasonable request.

REFERENCES:
- [Derived] Marruganti C, Romandini M, Gaeta C, Trovato E, Cinotti E, Rubegni P, D'Aiuto F, Grandini S. Treatment of periodontitis ameliorates the severity and extent of psoriasis-A randomized clinical trial. J Periodontal Res. 2025 Feb;60(2):134-143. doi: 10.1111/jre.13314. Epub 2024 Jun 20. PMID 38899599